CLINICAL TRIAL: NCT01998620
Title: Efficacy and Safety of S-adenosyl-L-methionine in Treatment of Chronic Hepatitis B Patients With Cholestasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMX-HBV-001
Record Dates: First submitted 2013-11-14; First posted 2013-12-02 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis B; Cholestasis
Keywords: Hepatitis B; Cholestasis
MeSH Terms: conditions — Hepatitis B; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ademetionine 1 (Experimental): Ademetionine 2000mg
  Interventions: Drug: Ademetionine 1
- Ademetionine 2 (Experimental): Ademetionine 1000mg
  Interventions: Drug: Ademetionine 2
- Ademetionine 3 (Active Comparator): no treatment in first 2 weeks, then Ademetionine 1000mg bid po with general antiviral treatment for 8 weeks
  Interventions: Drug: Ademetionine 3

INTERVENTIONS:
Drug: Ademetionine 2 — Ademetionine 1000mg ivgtt qd with general antiviral treatment for 2 weeks, then Ademetionine 500mg po bid with general antiviral treatment for 8 weeks
  Arms: Ademetionine 2
Drug: Ademetionine 1 — Ademetionine 2000mg ivgtt qd with general antiviral treatment for 2 weeks, then Ademetionine 1000mg bid po with general antiviral treatment for 8 weeks
  Arms: Ademetionine 1
Drug: Ademetionine 3 — no treatment for 2 weeks, then Ademetionine 1000mg bid po with general antiviral treatment for 8 weeks
  Arms: Ademetionine 3

SUMMARY:
This is an evaluation of adenosine methionine for treatment of chronic hepatitis b patients with cholestasis efficacy and safety of multicenter, randomized, open label clinical trial.

DETAILED DESCRIPTION:
evaluation of adenosine methionine for treatment of chronic hepatitis b patients with cholestasis efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. from 18-65 years old
2. diagnosed as hepatitis B, previous has HBV or HBsAg(+)>6 months, and now HBsAg or HBV DNA(+)
3. with intrahepatic cholestasis: meet EASL 2009 diagnoses criteria ALP>1.5ULN and GGT>3ULN or STB>2ULN

Exclusion Criteria:

1. liver mass, liver carcinoma
2. liver failure
3. non-hepatic diseases caused jaundice
4. obstructive jaundice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
levels of serum total bilirubin declined from baseline | 2 weeks
  levels of serum total bilirubin declined from baseline
Alkaline Phosphatase | 10 weeks
  Alkaline Phosphatase
Gamma-Glutamyl Transpeptidase | 10 weeks
  Gamma-Glutamyl Transpeptidase

SECONDARY OUTCOMES:
level of serum direct bilirubin decline from baseline | 2 weeks, 6 weeks, 10 weeks
  level of serum direct bilirubin decline from baseline
level of serum bile acids decline from baseline | 2 weeks, 6 weeks, 10 weeks
  level of serum bile acids decline from baseline
glutamic pyruvic transaminase | 2 weeks, 6 weeks, 10 weeks
  glutamic pyruvic transaminase
glutamic oxaloacetic transaminase | 2 weeks, 6 weeks, 10 weeks
  glutamic oxaloacetic transaminase

CONTACTS AND LOCATIONS:
Overall Officials: Liang Chen, Principal Investigator — Public Health Clinical Center Affiliated to Fudan University
Locations (1):
- Public Health Clinical Center Affiliated to Fudan University, Shanghai, Shanghai Municipality, China